CLINICAL TRIAL: NCT00615914
Title: Pramipexole Special Survey on Long-Term Use
Brief Title: Special Survey on Parkinson's Disease Patients Treated Long-term Use of Pramipexole
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.547
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The survey is conducted to collect safety and effectiveness information on the use of Pramipexole for long time of period in daily clinical settings in Japan.

ELIGIBILITY:
Inclusion Criteria:

Patients with Parkinson's disease

Exclusion Criteria:

Patients should have been treated according to the Japanese insert slip

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's disease patients in daily clinical settings
Sampling Method: Non-Probability Sample
Enrollment: 1645 (Actual)
Dates: Start 2004-02; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (272):
- Japan (272):
  - Boehringer Ingelheim Investigational Site, Agano
  - Boehringer Ingelheim Investigational Site, Aizu-Wakamatsu
  - Boehringer Ingelheim Investigational Site, Akashi
  - Boehringer Ingelheim Investigational Site, Akita
  - Boehringer Ingelheim Investigational Site, Asahikawa
  - Boehringer Ingelheim Investigational Site, Asakura
  - Boehringer Ingelheim Investigational Site, Azumino
  - Boehringer Ingelheim Investigational Site, Bandō
  - Boehringer Ingelheim Investigational Site, Beppu
  - Boehringer Ingelheim Investigational Site, Bihoro
  - Boehringer Ingelheim Investigational Site, Chiba
  - Boehringer Ingelheim Investigational Site, Chikusei
  - Boehringer Ingelheim Investigational Site, Chūō
  - Boehringer Ingelheim Investigational Site, Date
  - Boehringer Ingelheim Investigational Site, Ebetsu
  - Boehringer Ingelheim Investigational Site, Ebina
  - Boehringer Ingelheim Investigational Site, Fuchū
  - Boehringer Ingelheim Investigational Site, Fuji
  - Boehringer Ingelheim Investigational Site, Fujieda
  - Boehringer Ingelheim Investigational Site, Fujinomiya
  - Boehringer Ingelheim Investigational Site, Fujioka
  - Boehringer Ingelheim Investigational Site, Fujisawa
  - Boehringer Ingelheim Investigational Site, Fujiyoshida
  - Boehringer Ingelheim Investigational Site, Fukaya
  - Boehringer Ingelheim Investigational Site, Fukui
  - Boehringer Ingelheim Investigational Site, Fukuoka
  - Boehringer Ingelheim Investigational Site, Fukushima
  - Boehringer Ingelheim Investigational Site, Fukuyama
  - Boehringer Ingelheim Investigational Site, Gifu
  - Boehringer Ingelheim Investigational Site, Ginowan
  - Boehringer Ingelheim Investigational Site, Hachinohe
  - Boehringer Ingelheim Investigational Site, Hadano
  - Boehringer Ingelheim Investigational Site, Hagahama
  - Boehringer Ingelheim Investigational Site, Hakodate
  - Boehringer Ingelheim Investigational Site, Hamada
  - Boehringer Ingelheim Investigational Site, Hamamatsu
  - Boehringer Ingelheim Investigational Site, Hayashima
  - Boehringer Ingelheim Investigational Site, Higashimurayama
  - Boehringer Ingelheim Investigational Site, Higashiosaka
  - Boehringer Ingelheim Investigational Site, Higashiyamato
  - Boehringer Ingelheim Investigational Site, Himeji
  - Boehringer Ingelheim Investigational Site, Hiratsuka
  - Boehringer Ingelheim Investigational Site, Hirokawa
  - Boehringer Ingelheim Investigational Site, Hirosaki
  - Boehringer Ingelheim Investigational Site, Hiroshima
  - Boehringer Ingelheim Investigational Site, Hita
  - Boehringer Ingelheim Investigational Site, Hōfu
  - Boehringer Ingelheim Investigational Site, Ibaraki
  - Boehringer Ingelheim Investigational Site, Ichikikushikino
  - Boehringer Ingelheim Investigational Site, Ichinomiya
  - Boehringer Ingelheim Investigational Site, Ichinoseki
  - Boehringer Ingelheim Investigational Site, Iijima
  - Boehringer Ingelheim Investigational Site, Iizuka
  - Boehringer Ingelheim Investigational Site, Ikeda
  - Boehringer Ingelheim Investigational Site, Ikoma
  - Boehringer Ingelheim Investigational Site, Ina
  - Boehringer Ingelheim Investigational Site, Inazawa
  - Boehringer Ingelheim Investigational Site, Inba
  - Boehringer Ingelheim Investigational Site, Inuyama
  - Boehringer Ingelheim Investigational Site, Isesaki
  - Boehringer Ingelheim Investigational Site, Itoigawa
  - Boehringer Ingelheim Investigational Site, Iwaki
  - Boehringer Ingelheim Investigational Site, Iwata
  - Boehringer Ingelheim Investigational Site, Jōetsu
  - Boehringer Ingelheim Investigational Site, Kagoshima
  - Boehringer Ingelheim Investigational Site, Kahoku
  - Boehringer Ingelheim Investigational Site, Kajiki
  - Boehringer Ingelheim Investigational Site, Kakegawa
  - Boehringer Ingelheim Investigational Site, Kakogawa
  - Boehringer Ingelheim Investigational Site, Kamisu
  - Boehringer Ingelheim Investigational Site, Kamogawa
  - Boehringer Ingelheim Investigational Site, Kanazawa
  - Boehringer Ingelheim Investigational Site, Kanegusuku
  - Boehringer Ingelheim Investigational Site, Kannonji
  - Boehringer Ingelheim Investigational Site, Karatsu
  - Boehringer Ingelheim Investigational Site, Kashima
  - Boehringer Ingelheim Investigational Site, Kashiwa
  - Boehringer Ingelheim Investigational Site, Kashiwazaki
  - Boehringer Ingelheim Investigational Site, Kasukabe
  - Boehringer Ingelheim Investigational Site, Katō
  - Boehringer Ingelheim Investigational Site, Kawagoe
  - Boehringer Ingelheim Investigational Site, Kawasaki
  - Boehringer Ingelheim Investigational Site, Kawatana
  - Boehringer Ingelheim Investigational Site, Kikugawa
  - Boehringer Ingelheim Investigational Site, Kirishima
  - Boehringer Ingelheim Investigational Site, Kitakyushu
  - Boehringer Ingelheim Investigational Site, Kiyose
  - Boehringer Ingelheim Investigational Site, Kiyotake
  - Boehringer Ingelheim Investigational Site, Kizugawa
  - Boehringer Ingelheim Investigational Site, Kobayashi
  - Boehringer Ingelheim Investigational Site, Kobe
  - Boehringer Ingelheim Investigational Site, Kochi
  - Boehringer Ingelheim Investigational Site, Kodaira
  - Boehringer Ingelheim Investigational Site, Kofu
  - Boehringer Ingelheim Investigational Site, Koga
  - Boehringer Ingelheim Investigational Site, Kokubunji
  - Boehringer Ingelheim Investigational Site, Komae
  - Boehringer Ingelheim Investigational Site, Komatsu
  - Boehringer Ingelheim Investigational Site, Komoro
  - Boehringer Ingelheim Investigational Site, Koshikawa
  - Boehringer Ingelheim Investigational Site, Kōriyama
  - Boehringer Ingelheim Investigational Site, Kōshi
  - Boehringer Ingelheim Investigational Site, Kōtari
  - Boehringer Ingelheim Investigational Site, Kumamoto
  - Boehringer Ingelheim Investigational Site, Kurashiki
  - Boehringer Ingelheim Investigational Site, Kurayoshi
  - Boehringer Ingelheim Investigational Site, Kure
  - Boehringer Ingelheim Investigational Site, Kurume
  - Boehringer Ingelheim Investigational Site, Kushiro
  - Boehringer Ingelheim Investigational Site, Kutchan
  - Boehringer Ingelheim Investigational Site, Kuwana
  - Boehringer Ingelheim Investigational Site, Kyoto
  - Boehringer Ingelheim Investigational Site, Maebaru
  - Boehringer Ingelheim Investigational Site, Maebashi
  - Boehringer Ingelheim Investigational Site, Maibara
  - Boehringer Ingelheim Investigational Site, Maizuru
  - Boehringer Ingelheim Investigational Site, Marugame
  - Boehringer Ingelheim Investigational Site, Matsuda
  - Boehringer Ingelheim Investigational Site, Matsudo
  - Boehringer Ingelheim Investigational Site, Matsue
  - Boehringer Ingelheim Investigational Site, Matsumoto
  - Boehringer Ingelheim Investigational Site, Matsuyama
  - Boehringer Ingelheim Investigational Site, Mibu
  - Boehringer Ingelheim Investigational Site, Mihara
  - Boehringer Ingelheim Investigational Site, Miki
  - Boehringer Ingelheim Investigational Site, Minakami
  - Boehringer Ingelheim Investigational Site, Minamata
  - Boehringer Ingelheim Investigational Site, Minobu
  - Boehringer Ingelheim Investigational Site, Misashino
  - Boehringer Ingelheim Investigational Site, Mito
  - Boehringer Ingelheim Investigational Site, Miyaki
  - Boehringer Ingelheim Investigational Site, Miyakonojō
  - Boehringer Ingelheim Investigational Site, Miyazaki
  - Boehringer Ingelheim Investigational Site, Mooka
  - Boehringer Ingelheim Investigational Site, Moriguchi
  - Boehringer Ingelheim Investigational Site, Morioka
  - Boehringer Ingelheim Investigational Site, Moriya
  - Boehringer Ingelheim Investigational Site, Moriyama
  - Boehringer Ingelheim Investigational Site, Motona
  - Boehringer Ingelheim Investigational Site, Mukai-awagasaki
  - Boehringer Ingelheim Investigational Site, Muroran
  - Boehringer Ingelheim Investigational Site, Nagakute
  - Boehringer Ingelheim Investigational Site, Nagaoka
  - Boehringer Ingelheim Investigational Site, Nagasaki
  - Boehringer Ingelheim Investigational Site, Nagoya
  - Boehringer Ingelheim Investigational Site, Nangōku
  - Boehringer Ingelheim Investigational Site, Nara
  - Boehringer Ingelheim Investigational Site, Narita
  - Boehringer Ingelheim Investigational Site, Narutō
  - Boehringer Ingelheim Investigational Site, Nichinan
  - Boehringer Ingelheim Investigational Site, Niigata
  - Boehringer Ingelheim Investigational Site, Niihama
  - Boehringer Ingelheim Investigational Site, Nikkō
  - Boehringer Ingelheim Investigational Site, Nishigō
  - Boehringer Ingelheim Investigational Site, Nishihara
  - Boehringer Ingelheim Investigational Site, Nishinomiya
  - Boehringer Ingelheim Investigational Site, Nishio
  - Boehringer Ingelheim Investigational Site, Nishitōkyō
  - Boehringer Ingelheim Investigational Site, Nobeoka
  - Boehringer Ingelheim Investigational Site, Noboribetsu
  - Boehringer Ingelheim Investigational Site, Numazu
  - Boehringer Ingelheim Investigational Site, Obama
  - Boehringer Ingelheim Investigational Site, Obihiro
  - Boehringer Ingelheim Investigational Site, Odawara
  - Boehringer Ingelheim Investigational Site, Ohzu
  - Boehringer Ingelheim Investigational Site, Ojiya
  - Boehringer Ingelheim Investigational Site, Okayama
  - Boehringer Ingelheim Investigational Site, Omaezaki
  - Boehringer Ingelheim Investigational Site, Omuta
  - Boehringer Ingelheim Investigational Site, Onomichi
  - Boehringer Ingelheim Investigational Site, Osaka
  - Boehringer Ingelheim Investigational Site, Ōdate
  - Boehringer Ingelheim Investigational Site, Ōfunato
  - Boehringer Ingelheim Investigational Site, Ōgaki
  - Boehringer Ingelheim Investigational Site, Ōiso
  - Boehringer Ingelheim Investigational Site, Ōita
  - Boehringer Ingelheim Investigational Site, Ōkawa
  - Boehringer Ingelheim Investigational Site, Ōmura
  - Boehringer Ingelheim Investigational Site, Ōnojō
  - Boehringer Ingelheim Investigational Site, Ōtsu
  - Boehringer Ingelheim Investigational Site, Ōzu
  - Boehringer Ingelheim Investigational Site, Sado
  - Boehringer Ingelheim Investigational Site, Saga
  - Boehringer Ingelheim Investigational Site, Sagamihara
  - Boehringer Ingelheim Investigational Site, Saitama
  - Boehringer Ingelheim Investigational Site, Sakai
  - Boehringer Ingelheim Investigational Site, Sakaidechō
  - Boehringer Ingelheim Investigational Site, Sakata
  - Boehringer Ingelheim Investigational Site, Saku
  - Boehringer Ingelheim Investigational Site, Sanjō
  - Boehringer Ingelheim Investigational Site, Sano
  - Boehringer Ingelheim Investigational Site, Sanyōonoda
  - Boehringer Ingelheim Investigational Site, Sapporo
  - Boehringer Ingelheim Investigational Site, Sasebo
  - Boehringer Ingelheim Investigational Site, Seijō
  - Boehringer Ingelheim Investigational Site, Sendai
  - Boehringer Ingelheim Investigational Site, Shimabara
  - Boehringer Ingelheim Investigational Site, Shimonoseki
  - Boehringer Ingelheim Investigational Site, Shimotsuke
  - Boehringer Ingelheim Investigational Site, Shingū
  - Boehringer Ingelheim Investigational Site, Shinshiro
  - Boehringer Ingelheim Investigational Site, Shizuoka
  - Boehringer Ingelheim Investigational Site, Shūnan
  - Boehringer Ingelheim Investigational Site, Soo
  - Boehringer Ingelheim Investigational Site, Suita
  - Boehringer Ingelheim Investigational Site, Tajimi
  - Boehringer Ingelheim Investigational Site, Takamatsu
  - Boehringer Ingelheim Investigational Site, Takanabe
  - Boehringer Ingelheim Investigational Site, Takaoka
  - Boehringer Ingelheim Investigational Site, Takasago
  - Boehringer Ingelheim Investigational Site, Takasaki
  - Boehringer Ingelheim Investigational Site, Takatsuki
  - Boehringer Ingelheim Investigational Site, Takehara
  - Boehringer Ingelheim Investigational Site, Takinomiya
  - Boehringer Ingelheim Investigational Site, Toda
  - Boehringer Ingelheim Investigational Site, Togitsu
  - Boehringer Ingelheim Investigational Site, Tokoname
  - Boehringer Ingelheim Investigational Site, Tokushima
  - Boehringer Ingelheim Investigational Site, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Edogawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Katsushika-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Kita-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Minayo-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nakano-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Suginami-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site, Tomakomai
  - Boehringer Ingelheim Investigational Site, Tomiai
  - Boehringer Ingelheim Investigational Site, Tondabayashi
  - Boehringer Ingelheim Investigational Site, Toride
  - Boehringer Ingelheim Investigational Site, Toyama
  - Boehringer Ingelheim Investigational Site, Toyoake
  - Boehringer Ingelheim Investigational Site, Toyokawa
  - Boehringer Ingelheim Investigational Site, Toyonaka
  - Boehringer Ingelheim Investigational Site, Toyooka
  - Boehringer Ingelheim Investigational Site, Tōon
  - Boehringer Ingelheim Investigational Site, Tsu
  - Boehringer Ingelheim Investigational Site, Tsubata
  - Boehringer Ingelheim Investigational Site, Tsuchiura
  - Boehringer Ingelheim Investigational Site, Tsukuba
  - Boehringer Ingelheim Investigational Site, Tsuruoka
  - Boehringer Ingelheim Investigational Site, Ueda
  - Boehringer Ingelheim Investigational Site, Uji
  - Boehringer Ingelheim Investigational Site, Ujo
  - Boehringer Ingelheim Investigational Site, Urayasu
  - Boehringer Ingelheim Investigational Site, Uruma
  - Boehringer Ingelheim Investigational Site, Utsunomiya
  - Boehringer Ingelheim Investigational Site, Wajiki
  - Boehringer Ingelheim Investigational Site, Wakayama
  - Boehringer Ingelheim Investigational Site, Yamagata
  - Boehringer Ingelheim Investigational Site, Yamaguchi
  - Boehringer Ingelheim Investigational Site, Yamamoto
  - Boehringer Ingelheim Investigational Site, Yanai
  - Boehringer Ingelheim Investigational Site, Yao
  - Boehringer Ingelheim Investigational Site, Yashiro
  - Boehringer Ingelheim Investigational Site, Yazu
  - Boehringer Ingelheim Investigational Site, Yokkaichi
  - Boehringer Ingelheim Investigational Site, Yokohama
  - Boehringer Ingelheim Investigational Site, Yokote
  - Boehringer Ingelheim Investigational Site, Yoro
  - Boehringer Ingelheim Investigational Site, Yoshinogawa
  - Boehringer Ingelheim Investigational Site, Yufu
  - Boehringer Ingelheim Investigational Site, Zama

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: Pramipexole tablets - oral administration (0.125 mg and 0.5 mg)
Period: Overall Study
Arm/Group | Pramipexole
Started | 1645 (The number of patients enrolled)
Completed | 1008
Not Completed | 637
Not completed — Adverse Event | 274
Not completed — Death | 20
Not completed — Lack of Efficacy | 59
Not completed — Lost to Follow-up | 187
Not completed — Withdrawal by Subject | 16
Not completed — Physician Decision | 4
Not completed — No data was collected. | 65
Not completed — No treatment | 2
Not completed — Irregularly enrolled patients | 10

BASELINE CHARACTERISTICS:
Population: Data set for safety analysis - The number of patients enrolled was 1645. The number of case report forms which were collected was 1581. Moreover the number of patients analyzed as safety analysis was 1553 because 28 patients were excluded due to protocol violations.
Groups:
- Pramipexole: Pramipexole tablets were administered orally to patients according to the package insert in Japan. The drug form is only tablet. The initial dose was 0.125 mg twice a day, and was escalated until symptom control was achieved. The maintenance dose was between 1.5 mg/day and 4.5 mg/day (0.5 mg - 1.5 mg three times a day).
Arm/Group | Pramipexole
Number analyzed (Participants) | 1553
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 890
  Male | 663

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Global Impression of Improvement
Description: Investigators evaluation of the PD symptoms on a rating scale of 5 categories (very much improved, much improved, minimally improved, no effect, and unassessable).
Time Frame: 18 months
Population: A total of 26 patients were excluded from 1553 patients (Administration to patients who did not suffer from PD: 20, No efficacy data available: 6). As a result, 1527 patients included to the efficacy analysis set.
Measure: Number; unit: Participants
Groups:
- Pramipexole: The drug was administered orally to patients according to the package insert in Japan. The drug form is only tablet. The initial dose was 0.125 mg twice a day, and was escalated in case of lack of efficacy. The maintenance dose was between 1.5 mg/day and 4.5 mg/day (0.5 mg - 1.5 mg three times a day).
Arm/Group | Pramipexole
Number analyzed (Participants) | 1527
Participants
  Very much improved | 48
  Much improved | 561
  Minimally improved | 484
  No effect | 209
  Unassessable | 225

2. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score
Description: Motor examination is assessed by 27 questionnaire items in UPDRS Part III section. Each item is scored from 0 (best) to 4 (worst), and the total score of UPDRS Part III is from 0 (best) to 108 (worst). A decrease in the score means improvement.
Time Frame: Baseline and at 18 months (or at the time of discontinuation)
Population: The number of patients from the efficacy analysis set (1527) who had the assessment of UPDRS Part III total score at baseline and at or after 18 months of treatment or at the time of discontinuation (1356).
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 1356
Unit on a scale | -5.4 (10.7)

3. Secondary Outcome: Change From Baseline in Modified Hoehn & Yahr Rating Scale
Description: A severity of PD symptom are assessed by Modified Hoehn & Yahr rating scale. This scale consist of 10 levels including additional evaluation levels defined in Japan. Ten levels are described by 0 (best), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5 (worst).
Time Frame: Baseline and at 18 months (or at the time of discontinuation)
Population: The number of patients from the efficacy analysis set (1527) who had the assessment of Modified Hoehn & Yahr rating scale at baseline and at or after 18 months of treatment or at the time of discontinuation (1430).
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 1430
Unit on a scale | -0.2 (0.6)

4. Primary Outcome: Proportion of Adverse Events, Adverse Drug Reactions, Serious Adverse Events
Description: The aim of this Post Marketing Surveillance (PMS) was to obtain long-term safety data with treatment of pramipexole in Parkinson's disease (PD) patients. Therefore these items were considered as a safety evaluation.
Time Frame: during 18 months
Population: Patients excluded from 1581 patients were: 15 who had no visit since the first prescription, 2 for no treatment, 10 patients who were irregularly enrolled patients (exclusion from analysis according to regulatory requirement) and 1 patient that had no safety data available. As a result, there were 1553 patients in the safety analysis set.
Measure: Number; unit: percentage of participants
Groups:
- Pramipexole: Pramipexole tablets were administered orally to patients according to the package insert in Japan. The drug form is only tablet. The initial dose was 0.125 mg twice a day, and was escalated in case of lack of efficacy. The maintenance dose was between 1.5 mg/day and 4.5 mg/day (0.5 mg - 1.5 mg three times a day).
Arm/Group | Pramipexole
Number analyzed (Participants) | 1553
percentage of participants
  Proportion of Adverse Events | 42.4
  Proportion of Adverse Drug Reactions | 34.5
  Proportion of Serious Adverse Events | 7.2

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Pramipexole: Pramipexole tablets - oral administration (0.125 mg and 0.5 mg) was administered orally to patients according to the package insert in Japan. The drug form is only tablet. The initial dose was 0.125 mg twice a day, and was escalated in case of lack of efficacy. The maintenance dose was between 1.5 mg/day and 4.5 mg/day (0.5 mg - 1.5 mg three times a day).
Arm/Group | Pramipexole
Serious Adverse Events (participants affected / at risk) | 111/1553
Other Adverse Events (participants affected / at risk) | 267/1553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramipexole (N=1553)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 16 (16)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pyothorax (Infections and infestations) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 3 (3)
Delirium (Psychiatric disorders) | 7 (7)
Delusion (Psychiatric disorders) | 6 (6)
Hallucination (Psychiatric disorders) | 7 (7)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Persecutory delusion (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2)
Coma hepatic (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Sudden onset of sleep (Nervous system disorders) | 3 (3)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Putamen haemorrhage (Nervous system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Shock (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Crush syndrome (Renal and urinary disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Drowning (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (8)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (4)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramipexole (N=1553)
Hallucination (Psychiatric disorders) | 131 (131)
Somnolence (Nervous system disorders) | 148 (148)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.